CLINICAL TRIAL: NCT04346771
Title: The Effect of Emotional Working Memory Training on Reducing Depressive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Wenhui Yang, Department of Psychology, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMOTION 2019
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Depressive Symptoms
Keywords: Depression; Cognitive control; Emotion; Working memory; Cognitive bias; Emotional regulation
MeSH Terms: conditions — Depression; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maintaining Positive Working memory (Experimental): Maintaining positive working memory training is based on visual positive works n-back task.In this training, positive words are presented on the pictures of happy face.According to the rules, subjects are required to identify whether the word present currently is as the same type as the word presented n before then click the keys correspondingly.Each training session contains 15 blocks which are consisted with 20+n trails.
  Interventions: Behavioral: Working memory training
- Positive Attention Bias Modification (Placebo Comparator): In the positive attention bias, there are 54 pairs of neutral-negative words, 27 pairs of which are used in the training group and 27 pairs of which are used in the placebo group. The word pairs in each group are repeated 8 times, with a total of 216 trial.Participants received 10 sessions over 2 weeks. 90% of the targets in the training group appear in the positive word position and 10% of the targets appear in the neutral word position.
  Interventions: Behavioral: Positive ABMT

INTERVENTIONS:
Behavioral: Working memory training — Participants complete 10 sessions of maintaining positive working memory training during a two-week period. Each session consists of 15 blocks.
  Arms: Maintaining Positive Working memory
Behavioral: Positive ABMT — Participants complete 8 sessions of attention bias modification training (ABMT) during a two-week period. Each session consists of 218 trials, and the time to complete a training session is 12 minutes.
  Arms: Positive Attention Bias Modification

SUMMARY:
The purpose of this study is to test whether emotional working memory training and attention bias modification training are an effective neurobehavioral therapy to improve depressive symptoms.That is whether emotional working memory training is superior to attention bias modification training or not in reducing depressive symptoms over 1 year after training.

DETAILED DESCRIPTION:
Attentional bias has been theorized to play a critical role in the onset and maintenance of depression. Attentional bias modification training (ABMT), an experimental paradigm that uses training to induce adaptive attentional bias, was developed to test the causal model and this has therapeutic implications in depression.To test the effect of ABMT on treatment of depressive symptoms, a randomized, double-blind, placebo and blank controlled trial is conducted in college students who are experiencing mild-to-severe symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

Meet the major and mild depression disorder's criteria

Exclusion Criteria:

bipolar disorder, schizophrenia or organic mental disorder; any concurrent psychotherapy; any concurrent psychotropic medication.

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-01-10 (Estimated); Study Completion 2021-01-10 (Estimated)

PRIMARY OUTCOMES:
Changes of depressive symptoms | pre-training, post-training(2 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month( booster pre-training), 4-month (booster post-training), 5-month,6-month,12-month after post-training)
  Depression symptoms tested by clinicians using the Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS)

SECONDARY OUTCOMES:
Changes of self-reported depressive symptoms | pre-training, post-training(2 weeks after pre-training), follow-ups(1-week,2-week,4-week,7-week,3-month( booster pre-training), 4-month (booster post-training), 5-month,6-month,12-month after post-training)
  Self-reported depressive symptoms assessed by Beck depression scale-second version (BDI-II)

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Yang, Principal Investigator — Department of Psychology, Hunan Normal University
Locations (1):
- Department of Psychology, Hunan Normal University, Changsha, Hunan, China